CLINICAL TRIAL: NCT06555302
Title: Cognitive Priming to Boost Stroke Tele-rehabilitation Outcomes
Brief Title: Cognitive Priming for Stroke Tele-rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Stephanie Aghamoosa, Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00136303; 3P20GM109040-10S2 (NIH)
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Cognitive Training; Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Rehabilitation + Occupational Therapy (Telerehabilitation) (Experimental): A trained OT will deliver the 8-week stroke telerehabilitation program. There will be 13 total sessions with 2 sessions/week for the first 5 weeks and 1 session/week for the last 3 weeks. The cognitive rehabilitation and OT components will be titrated as follows:
  * Sessions 1-4 will focus on cognitive rehab.
  * Sessions 5-10 will review/provide additional cognitive rehab and deliver OT.
  * Sessions 11-13 may briefly review cognitive rehab but focus primarily on OT.
  Interventions: Behavioral: Cognitive Rehabilitation; Behavioral: Occupational Therapy

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation — Cognitive rehabilitation will be OT-led, one-on-one sessions focused on teaching cognitive strategies and their application to a broad set of activities/settings. The goal is to facilitate cognitive skill learning and generalization, by applying the new cognitive strategies to the participant's performance of home-based and community-based activities (taught through the subsequent OT portion of the intervention).
Behavioral: Occupational Therapy — OT upper extremity rehabilitation will have 2 components: task-practice and metacognitive strategy training. The task-practice involves a patient repetitively practicing stroke-impaired movement skills within the context of a functional task to promote recovery of the impaired skills. THE task practice sessions will be coached/guided by the therapist through a metacognitive strategy training process which is based on the Cognitive Orientation to Occupational Performance (CO-OP) approach aimed at enhancing self-management during home and community living tasks.

SUMMARY:
The goal of this pilot study is to investigate whether adding cognitive rehabilitation to an existing occupational therapy (OT) stroke telerehabilitation program will improve stroke survivors' functioning. The main question it aims to answer is whether this intervention improves cognition, participation, upper extremity use in real-world activities, and mood/quality of life. Participants will be asked to engage in an 8-week stroke tele-rehabilitation program (13 sessions), which includes both cognitive rehabilitation and OT for arm/hand function, and complete assessments before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Have experienced ischemic or hemorrhagic stroke with resultant paresis of one arm/hand at least 30 days prior
* Adults ages 21 years or older
* Are able to speak and read English
* Have corrected vision to be able to read text on a screen
* Have a device on which a telerehabilitation visit can be conducted (i.e., phone, tablet, or laptop) and a Wi-Fi connection or cellular service
* Able to participate in the study's assessment sessions as per the judgment of the licensed, experienced stroke telerehabilitation occupational therapist.

Exclusion Criteria:

* Have moderate-severe or severe aphasia.
* Have impaired decision making capacity as determined by a standard protocol for assessing capacity to provide informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Change From Baseline Global Cognition, as Measured by the Montreal Cognitive Assessment (MoCA) | Baseline prior to treatment and at post-assessment within 10 days post-treatment
  Montreal Cognitive Assessment (MoCA) is a 16-item objective cognitive screening measure. The maximum possible score = 30 points with higher scores indicating better cognition. Any necessary modifications for remote administration will be made according to guidelines provided on the official MoCA website (https://mocacognition.com/remote-moca-testing/).
Change From Baseline Functional Task Performance and Activity Participation, as Measured by the Patient Specific Functional Scale (PSFS) | Baseline prior to treatment and at post-assessment within 10 days post-treatment
  Patient Specific Functional Scale (PSFS) is a patient-reported measure of task-goal identification and difficulty performing the task on a 0-10-point ordinal scale with higher ratings indicating greater satisfaction with task performance.
Change From Baseline Psychosocial Function (Depression), as Measured by the Patient Health Questionnaire (PHQ-9) | Baseline prior to treatment and at post-assessment within 10 days post-treatment
  Patient Health Questionnaire (PHQ-9) is a 9-item self-report measure of depression. Items query mood (feeling down, lack of interest), thoughts (guilt, suicidality), and physical symptoms (appetite, sleep, fatigue, concentration, restlessness). Each item is scored on a 4-point scale reflecting how often the symptom has occurred over the last 2 weeks (0=not at all, 3=nearly every day). Scores are summed (out of 27), with higher scores indicating more symptoms of depression.

SECONDARY OUTCOMES:
Change From Baseline Subjective Cognition, as Measured by the NeuroQoL-Cognitive Function | Baseline prior to treatment and at post-assessment within 10 days post-treatment
  NeuroQoL-Cognitive Function Short Form v.2.0 is a 29-item subjective measure of cognitive function. This patient-reported outcome assesses perceived abilities in memory, attention, decision making, or in the application of such abilities to everyday tasks (e.g., planning, organizing, calculating, remembering, and learning) on a 5-item rating scale (1=cannot do to 5=no difficulty). The summed raw score is converted into a normed T-score (mean=50, SD=10). Higher T-scores reflect better perceived cognitive function.
Change From Baseline Functional Task Performance and Activity Participation, as Measured by the Performance Quality Rating Scale (PQRS) | From intervention session #5 to intervention session #13 (5 weeks)
  Performance Quality Rating Scale (PQRS) is a therapist-rated measure. The OT observes the participant's performance of a task and rates it on a 0-10-point ordinal scale with higher ratings indicating greater task performance skill.
Change From Baseline Functional Task Performance and Activity Participation, as Measured by the Stroke Self Efficacy Questionnaire (SSEQ) | Baseline prior to treatment and at post-assessment within 10 days post-treatment
  Stroke Self Efficacy Questionnaire (SSEQ) is a 13-item self-report measure of confidence (0-10-point Likert scale with higher numbers indicating greater confidence) doing at-home tasks such as using both hands to eat food or prepare a meal for oneself.
Change From Baseline Psychosocial Function (Global), as Measured by the Inventory of Psychosocial Functioning | Baseline prior to treatment and at post-assessment within 10 days post-treatment
  Inventory of Psychosocial Functioning is an 80-item self-report measure of impairment in 7 psychosocial domains within the last 30 days: romantic relationships, family other than spouse/partner, work, friendships and socializing, parenting, education, and self-care. Participants rate the frequency of difficulty on each item on a 7-point scale (0=never, 6=always). Scores are averaged by domain and multiplied by 100; an overall score is the average of domain scores; higher scores indicate greater impairment in psychosocial function.
Change From Baseline Psychosocial Function (Sleep), as Measured by the PROMIS Sleep Disturbance | Baseline prior to treatment and at post-assessment within 10 days post-treatment
  PROMIS Sleep Disturbance is an 8-item self-report measure of perceived difficulties falling and/or staying asleep. Items are rated on a 5-point rating scale (1=no problem, 5=very much a problem). The summed raw score is converted into a normed T-score (mean=50, SD=10). Higher T-scores reflect more sleep disturbance.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared in the NIH-funded Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (DASH).

DOCUMENTS (1):
  • Informed Consent Form (2024-10-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT06555302/ICF_000.pdf